CLINICAL TRIAL: NCT00036140
Title: Study of the Safety and Efficacy of an Investigational Drug in Adult Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Purpose: Treatment
Other Study IDs: 196-ONC-0100-006
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-03

CONDITIONS: Multiple Myeloma
Keywords: Pharmacia
MeSH Terms: conditions — Multiple Myeloma | interventions — Drugs, Investigational

INTERVENTIONS:
Drug: Investigational drug

SUMMARY:
The primary goal of the study is to determine the best dose of an investigational drug to give to patients with multiple myeloma and to evaluate the investigational drug's effectiveness as a treatment for multiple myeloma.

ELIGIBILITY:
Other specific inclusion/exclusion criteria may apply. In order to determine eligibility, further examination by the investigator is necessary.

Inclusion Criteria:

* Eligible patients must be at least 18 years of age with a diagnosis of multiple myeloma including elevated M-blood/urine protein or a tumor that can be evaluated by the doctor during the investigational drug's treatment.
* The patient's multiple myeloma must have gotten worse during/after previous chemotherapy was given.
* Any side-effects from prior chemotherapy must have subsided
* Blood and urine tests must show adequate bone marrow, liver, and kidney function.

Exclusion Criteria:

Any of the following will exclude patients from study participation:

* indolent or smoldering myeloma or localized plasmacytoma
* hyperviscosity syndrome
* irradiation to 25% or more of bone marrow
* prior high dose chemotherapy with bone marrow or stem cell support
* current participation in other clinical trials
* pregnant or breast-feeding women
* known HIV-positive or AIDS-related illness
* patients planning to have radiation therapy or surgery that would interrupt study therapy in the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Center, Los Angeles, California
  - Research Center, Rancho Mirage, California
  - Research Center, Cleveland, Ohio
  - Research Center, Marshfield, Wisconsin